CLINICAL TRIAL: NCT04668365
Title: A Single Arm, Multi-center, Phase II Clinical Trial of Zanubrutinib Combined With Standard Chemotherapy in the Treatment for Patients With Diffuse Large B Cell Lymphoma and CD79A/CD79B Genetic Abnormality
Brief Title: Zanubrutinib Combined With Standard Chemotherapy in the Treatment for Patients With Diffuse Large B Cell Lymphoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Data in analysis
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhihua Yao, PhD, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYNHL05
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B Cell Lymphoma; CD79A Gene Mutation; CD79B Gene Mutation
Keywords: Diffuse Large B Cell Lymphoma; Zanubrutinib; CD79A/CD79B; Genetic Abnormality
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Congenital Abnormalities | interventions — Rituximab; zanubrutinib; Cyclophosphamide; Epirubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanubrutinib Combined With Standard Chemotherapy (Experimental): A: For the first-line treatment:
  Rituximab, 375mg/m2, Intravenous administration on day 0, combined with regimen：CHOP (Cyclophosphamide, Epirubicin, Vincristine and Prednisone): repeated every 3 weeks, up to 6 cycles.
  Zanubrutinib, 160mg twice daily continuous oral administration from 2 to 6 cycles for patients with CD79A/CD79B genetic abnormality.
  Zanubrutinib combined with Rituximab for the 7 cycle.
  B: For R/R DBCLC:
  Rituximab, 375mg/m2, Intravenous administration on day 0, combined with regimen: GemOx(Gemcitabine, Oxaliplatin)/ DHAP(Cisplatin, Cytarabine, Dexamethasone)/ ICE(Ifosfamide, Etoposide, Carboplatin)/ GDP(Gemcitabine, Cisplatin, Dexamethasone): repeated every 3 weeks, up to 5 cycles.
  Zanubrutinib, 160mg twice daily continuous oral administration from 2 to 5 cycles for patients with CD79A/CD79B genetic abnormality.
  Maintenance treatment: Zanubrutinib, 160mg twice daily continuous oral administration for 12 months.
  Interventions: Drug: Rituximab; Drug: Zanubrutinib; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — 375mg/m2, Intravenous administration on day 0 of each 3-week cycle.
  Other Names: RiTUXimab Injection
Drug: Zanubrutinib — 160mg twice daily continuous oral administration.
  Other Names: Zanubrutinib Pill
Drug: Cyclophosphamide — 750mg/m2, Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease after 2 cycles treatment, disease progression after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Cyclophosphamide Injection
Drug: Epirubicin — 70mg/m2, Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease after 2 cycles treatment, disease progression after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Epirubicin Injection
Drug: Vincristine — 1.4mg/m2 (Max: 2mg), Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease after 2 cycles treatment, disease progression after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Vincristine Injection
Drug: Prednisone — 100mg, oral administration on day 1 to 5 of each 3-week cycle until disease progression/stable disease after 2 cycles treatment, disease progression after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Prednisone Pill

SUMMARY:
This is a prospective single arm, multi-center, phase II clinical trial to observe the efficacy and safety of zanubrutinib combined with standard chemotherapy in the treatment for patients with diffuse large B cell lymphoma and CD79A/CD79B genetic abnormality.

DETAILED DESCRIPTION:
Diffuse large B cell lymphoma (DLBCL) is the most common type of non-Hodgkin's lymphoma (NHL). Currently, R-CHOP is world-widely used in the first-line treatment for DLBCL. There are about one second of patients suffering relapse and drug resistance. ABC-DLBCL mainly relies on the chronical activity of BCR signal, which can activate the downstream NF-kB pathway through BTK and MYD88, thereby promoting the occurrence of tumors. A study by Wyndham H Wilson et al. showed that 23% of ABC-DLBCL patients were accompanied by acquired functional mutations of the BCR component CD79A/CD79B. Zanubrutinib is a new BTK inhibitor. The goal of our trial is to assess the efficacy and safety of zanubrutinib combined with standard chemotherapy in the treatment for patients with diffuse large B cell lymphoma and CD79A/CD79B genetic abnormality.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old (including 18 and 75)
2. Diagnosed as diffuse large B cell lymphoma
3. CD79A/CD79B genetic abnormality
4. Subjects with untreated or relapsed/refractory DLBCL
5. Having at least one measurable lesions
6. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-1
7. Life expectancy no less than 3 months
8. enough main organ function
9. Pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and six months after this study
10. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Diagnosed as high-grade B-cell lymphoma, including non-specified and double-strike or triple-strike
2. Diagnosed as grey-zone lymphoma
3. Diagnosed as primary mediastinal large B-cell lymphoma
4. Diagnosed as CD20 negative diffuse large B-cell lymphoma
5. Active malignant tumor need be treated at the same time
6. Other malignant tumor history
7. Serious surgery and trauma less than two weeks
8. Systemic therapy for serious acute/chronic infection
9. Congestive heart failure, uncontrolled coronary heart disease, arrhythmia and heart infarction less than 6 months
10. Vaccination with live attenuated vaccine less than 4 weeks
11. HIV-positive, AIDS patients and untreated active hepatitis
12. Patients with a history of deep vein thrombosis or pulmonary embolism less than 12 months
13. Patients with a history of mental illness
14. Researchers determine unsuited to participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2020-12-25 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of complete remission for 3-4 weeks after induction treatment | from the date of the first cycle of treatment to 3-4 weeks after induction treatment of the last included patient (each cycle is 21 days)
  the total proportion of patients with complete remission (CR) for 3-4 weeks after induction treatment

SECONDARY OUTCOMES:
objective response rate | every 6 weeks from the day of the first cycle of induction chemotherapy treatment and every 8 weeks from the day of the first cycle of maintenance treatment to 18 months after last patient's enrollment (each cycle is 21 days)
  the total proportion of patients with complete response (CR) and partial response (PR)
2-year progression-free survival | from the day of the first cycle of treatment to the date of confirmed progressive disease or death, whichever occurs first, up to 2 years after last patient's enrollment (each cycle is 21 days)
  the total proportion of patients with no progression from date of the first day of treatment to the date of confirmed progressive disease or death which one occurs first
2-year overall survival | from date of the first cycle of treatment to the date of death from any cause, assessed up to 2 years (each cycle is 21 days)
  from date of first day of treatment to the date of death by any cause
incidence and relationship with study drugs of grade 3-4 adverse events | from the date of the first cycle of treatment to 18 months after last patient's enrollment (each cycle is 21 days)
  the incidence and relationship with study drugs of grade 3 or 4 adverse events (based on NCI CTC-AE v4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Yao, M.D. Ph.D, Study Director — Henan Cancer Hospital; Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China